CLINICAL TRIAL: NCT01358604
Title: ROR1 as a Novel Target for Neuroblastoma
Brief Title: Biomarkers in Samples From Young Patients With Neuroblastoma
Status: Completed | Type: Observational
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: ANBL11B2; COG-ANBL11B2 (Other: Children's Oncology Group); NCI-2011-02855 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); ANBL11B2 (Other: Children's Oncology Group)
Record Dates: First submitted 2011-05-18; First posted 2011-05-23 (Estimated); Last update posted 2016-04-15 (Estimated); Status verified 2016-04

CONDITIONS: Neuroblastoma
Keywords: localized resectable neuroblastoma; recurrent neuroblastoma; regional neuroblastoma; stage 4S neuroblastoma; localized unresectable neuroblastoma
MeSH Terms: conditions — Neuroblastoma | interventions — Polymerase Chain Reaction; Blotting, Western; Flow Cytometry; Immunohistochemistry

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Genetic: polymerase chain reaction
Genetic: protein expression analysis
Genetic: western blotting
Other: flow cytometry
Other: immunohistochemistry staining method
Other: laboratory biomarker analysis

SUMMARY:
RATIONALE: Studying samples of tissue and bone marrow from patients with cancer in the laboratory may help doctors learn more about changes that occur in DNA and identify biomarkers related to cancer.

PURPOSE: This research study studies biomarkers in samples from young patients with neuroblastoma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To analyze the expression of ROR1 on the surface of primary neuroblastoma cells.
* To investigate the therapeutic potential of anti-ROR1 monoclonal antibodies (mAbs), bispecific antibodies, and immunotoxins in in vitro and in vivo models of neuroblastoma.

OUTLINE: Archived bone marrow and tumor tissue samples are analyzed for ROR1 expression by flow cytometry, western blotting, qPCR, and IHC.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosed with neuroblastoma

  * With or without N-myc amplification
* Primary tumor samples as frozen tissue in liquid nitrogen or -80 degrees C
* Bone marrow samples from high-risk patients as peripheral blood mononuclear cells (PBMC) that have been cryopreserved with DMSO as viable cells to be used for flow cytometry or slides of bone marrow that can be used for immunohistochemistry

PATIENT CHARACTERISTICS:

* Not specified

PRIOR CONCURRENT THERAPY:

* Not specified

Max Age: 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients diagnosed with neuroblastoma.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2011-05; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
ROR1 is expressed on the surface of neuroblastoma cells and constitutes a suitable target for mAb therapy

CONTACTS AND LOCATIONS:
Overall Officials: David Hema, MD, MPH, Principal Investigator — NCI - Experimental Transplantation and Immunology Branch